CLINICAL TRIAL: NCT05747664
Title: An Open-label, Multi-center, Parallel, Single Oral Dose Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of DWP16001 in Subjects With Hepatic Impairment Compared With Subjects With Normal Hepatic Function
Brief Title: To Compare the Safety and PK/PD Characteristics of Subjects With Between Hepatic Impairment and Normal Hepatic Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_DWP16001110
Record Dates: First submitted 2023-02-08; First posted 2023-02-28 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DWP16001 to normal haptic function (Experimental): Normal hepatic function
  Interventions: Drug: DWP16001
- DWP16001 to Child-Pugh Class A (Experimental): Child-Pugh Class A
  Interventions: Drug: DWP16001
- DWP16001 to Child-Pugh Class B (Experimental): Child-Pugh Class B
  Interventions: Drug: DWP16001

INTERVENTIONS:
Drug: DWP16001 — 0.3mg
  Other Names: DWP16001 0.3mg

SUMMARY:
This study aims to evaluate the pharmacokinetics, pharmacodynamics, safety, and tolerability of DWP16001 in subjects with hepatic impairment compared with subjects with normal hepatic function.

DETAILED DESCRIPTION:
The study design is An open-label, multi-center, parallel, single oral dose study.

ELIGIBILITY:
Inclusion Criteria:

1. A person who has decided to participate voluntarily and agreed in writing prior to the screening procedure after understanding the detailed explanation of this clinical trial.
2. A person who is 19 years of age or more and under 80 years of age at the time of screening.
3. Those with a weight of 45.0 kg or more and 90.0 kg or less and a body mass index (BMI) of 18.0 kg/m2 or more and 30.0 kg/m2 or less.

Exclusion Criteria:

1. A person who has a history of gastrointestinal diseases (e.g., ulcer, inflammatory bowel disease, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (except simple appendectomy or hernia surgery) that may affect the absorption of DWP16001.
2. Those who are hypersensitive to drugs and other drugs (aspirin, antibiotics, etc.) including the SGLT2 inhibitor family or who have a history of clinically significant hypersensitivity reaction.
3. Serum Cr >1.5mg/dL or eGFR (CKD-EPI Cr) <60mL/min/1.73m2
4. Those who have used SGLT2 inhibitor family drugs within two weeks of the scheduled date of administration of DWP16001.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Cmax of DWP16001 | 0 to 48 hours
  Cmax of DWP16001
AUClast of DWP16001 | 0 to 48 hours
  AUClast of DWP16001

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea